CLINICAL TRIAL: NCT07350213
Title: Step-Aerobics Versus Core Exercise for Non-HDL Cholesterol Reduction in Sedentary Women With Overweight/Obesity
Brief Title: Step-Aerobics Versus Core Exercise for Non-HDL Cholesterol Reduction in Sedentary Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, OGUZHAN CELIK, ASSOCIATE PROFESSOR, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: muglaSKU2-C-OC-01
Record Dates: First submitted 2025-12-28; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Cholesterol (Total and HDL); Exercise
Keywords: Exercise; Overweight; Obesity; Women; Cholesterol, Non-HDL
MeSH Terms: conditions — Motor Activity; Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Two groups with a step aerobics group or a core exercise group
Who Masked: Investigator
Masking Description: The patients were randomly assigned, in a 1:1 ratio, into one of two groups of intervention: step-aerobics group (SAG) or core exercise group (CEG). An independent researcher produced the random sequence by computer-based random number generator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- step-aerobics group (Active Comparator): The aerobic-step exercise training protocol included methodically planned 60-minute training sessions with the following components:
  Warm-up Phase (10 minutes): Low-intensity aerobic movements that are intended to slowly raise heart rate and ready the cardiovascular system for more vigorous exercise. This phase consisted of low stepping movements, arm circles, and dynamic stretching exercises. Main Exercise Phase (40 minutes): Aerobic-step exercise routines done on adjustable step platforms.Step height was individualized according to participant fitness level and progressed incrementally during the course of the intervention. Exercises consisted of simple step-ups, lateral steps, knee lifts, and complex choreographed movement patterns incorporating both lower and upper body movements. Music with suitable tempo was used to help maintain rhythm and motivation. Cool-down Phase (10 minutes): Progressive decrease in the intensity of exercise coupled
  Interventions: Other: Step-Aerobics Group; Other: Core Exercise Group
- core exercise group (Active Comparator): Warm-up Phase (10 minutes): Simple aerobic movements akin to the step group but with focus on core engagement and spinal mobility. This phase involved marching in place, slow torso rotations, and preparatory core engagement exercises. Main Exercise Phase (40 minutes): Strength and stability exercises targeting the core and integrating aerobic movements. Planks, modified crunches, bridge exercises, stability ball exercises, Pilates160 inspired movements, and functional core strengthening exercises were included in this phase. The aerobic element was preserved by using continuous movement patterns and circuit-style training to keep heart rate within the desired zone.
  Interventions: Other: Step-Aerobics Group; Other: Core Exercise Group

INTERVENTIONS:
Other: Step-Aerobics Group — Step Aerobics: The primary goal is to improve cardiovascular health and burn calories. It mainly targets the lower body muscles, including the legs, glutes, and calves. The arms and core also engage to keep pace with the rhythm.
Other: Core Exercise Group — The primary goal is to stabilize and strengthen the body's center (abs, lower back, hips, and the area surrounding the spine). The focus is on resistance and balance rather than mobility. These exercises target the core region, including deep abdominal muscles, lower back muscles, the pelvic floor, and the diaphragm. They are generally more static (stationary) or controlled.

SUMMARY:
This study investigated the effects of a step-aerobics program versus a core exercise program on serum non-HDL-C levels and other cardiometabolic parameters in sedentary women with overweight/obesity.

DETAILED DESCRIPTION:
Non-high-density lipoprotein cholesterol (non-HDL-C) is a key predictor of cardiovascular disease (CVD), yet the comparative effects of different exercise modalities on this marker, particularly in high-risk populations, are not fully understood.

This study investigated the effects of a step-aerobics program versus a core exercise program on serum non-HDL-C levels and other cardiometabolic parameters in sedentary women with overweight/obesity.

Forty-five with overweight/obesity sedentary women were randomly assigned to either a step aerobics group (SAG; n=25) or a core exercise group (CEG; n=20). Both groups participated in supervised exercise sessions for 60 minutes, 4 days per week, for 16 weeks. Exercise intensity was prescribed and progressively increased from 60% to 70% of the heart rate reserve (HRR), determined by the Karvonen formula.

A 16-week supervised step-aerobics program is an effective intervention for improving the atherogenic lipid profile, particularly non-high-density lipoprotein cholesterol, in sedentary women with overweight or obesity.

ELIGIBILITY:
Inclusion Criteria:

* Female sex, aged 25-45 years.
* Sedentary lifestyle, defined as engaging in less than 150 minutes of moderate-intensity physical activity per week for the preceding six months.
* Overweight or Class I Obesity, defined according to World Health Organization (WHO) criteria as a Body Mass Index (BMI) between 25.0 and 34.9 kg/m².
* Willingness to participate in a 16-week supervised exercise program and provide written informed consent.

Exclusion Criteria:

* Presence of diagnosed CVD, uncontrolled hypertension (Systolic Blood Pressure >140 mmHg or Diastolic Blood Pressure >90 mmHg), or diabetes mellitus (Type 1 or 2).
* Current or past use (within 6 months) of lipid-lowering medications, antihypertensive drugs, or any medication known to affect metabolism.
* Active smoking.
* Pregnancy or lactation.
* Any musculoskeletal, orthopedic, or other medical condition that would prevent safe participation in the exercise programs.
* Participation in any structured, regular exercise program within the past six months.

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study investigated the effects of a step-aerobics program versus a core exercise program on serum non-HDL-C levels and other cardiometabolic parameters in sedentary women with overweight/obesity.
Enrollment: 45 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Serum Non-High-Density Lipoprotein Cholesterol (Non-HDL-C) levels measured via enzymatic assay (mg/dL)on HDL levels in overweight or obese, sedentary individuals. | Baseline (Week 0) and Post-Intervention (Week 16)
  Fasting venous blood samples will be collected at baseline and after the 16-week intervention. Serum Non-HDL-C will be calculated as Total Cholesterol minus High-Density Lipoprotein Cholesterol (HDL-C) using enzymatic assay methodology. Results will be reported as mean ± standard deviation (SD) and percentage change (%) from baseline. Between-group differences in change scores will be compared using independent samples t-tests with significance level set at p < 0.05.

SECONDARY OUTCOMES:
Serum Total Cholesterol levels measured via enzymatic assay (mg/dL) | Baseline (Week 0) and Post-Intervention (Week 16)
  Fasting venous blood samples will be collected at baseline and week 16. Total serum cholesterol will be measured using enzymatic assay. Data will be reported as mean ± SD and percentage change (%) from baseline. Bonferroni correction will be applied for multiple comparisons (adjusted α = 0.05/10).
Serum Low-Density Lipoprotein Cholesterol (LDL-C) levels measured via enzymatic assay (mg/dL) | Baseline (Week 0) and Post-Intervention (Week 16)
  Fasting venous blood samples will be collected at baseline and week 16. LDL-C will be measured using enzymatic assay. Results will be reported as mean ± SD and percentage change (%) from baseline. Statistical significance will be assessed using independent samples t-tests with Bonferroni correction applied (adjusted α = 0.05/10).
Serum High-Density Lipoprotein Cholesterol (HDL-C) levels measured via enzymatic assay (mg/dL) | Baseline (Week 0) and Post-Intervention (Week 16)
  Fasting venous blood samples will be collected at baseline and week 16. HDL-C will be measured using enzymatic assay. Data will be reported as mean ± SD and percentage change (%) from baseline. Between-group comparisons will be performed using independent samples t-tests with Bonferroni correction (adjusted α = 0.05/10).
Serum Triglycerides levels measured via enzymatic assay (mg/dL) | Baseline (Week 0) and Post-Intervention (Week 16)
  Fasting venous blood samples will be collected at baseline and week 16. Triglycerides will be measured using enzymatic assay. Results will be reported as mean ± SD and percentage change (%) from baseline. Statistical analysis will include independent samples t-tests with Bonferroni correction applied (adjusted α = 0.05/10).

OTHER OUTCOMES:
Body Mass Index (BMI) calculated from body weight and height (kg/m²) | Baseline (Week 0) and Post-Intervention (Week 16)
  Body weight (kg) and height (cm) will be measured at baseline and week 16 using calibrated scales and stadiometers. BMI will be calculated as weight (kg) divided by height (m²). Results will be reported as mean ± SD and absolute change from baseline. Between-group comparisons will be performed using independent samples t-tests.
Waist Circumference measured at the midpoint between the iliac crest and the lowest rib (cm) | Baseline (Week 0) and Post-Intervention (Week 16)
  Waist circumference will be measured at baseline and week 16 using a non-stretchable measuring tape positioned at the midpoint between the iliac crest and the lowest rib margin, with participants standing upright. Measurements will be recorded to the nearest 0.1 cm. Data will be reported as mean ± SD and absolute change from baseline. Statistical analysis will include independent samples t-tests for between-group comparisons.
Resting Heart Rate measured via validated heart rate monitors (beats per minute, bpm) | Baseline (Week 0) and Post-Intervention (Week 16)
  Resting heart rate will be measured at baseline and week 16 after participants have rested in a supine position for at least 5 minutes. Heart rate will be measured using validated heart rate monitors (Polar, Finland) placed on the chest. Results will be reported as mean ± SD and absolute change from baseline. Between-group differences will be compared using independent samples t-tests.

CONTACTS AND LOCATIONS:
Locations (1):
- Mugla Sitki Kocman University, Menteşe, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No